CLINICAL TRIAL: NCT01947309
Title: A Non-interventional, Observational Post-marketing Registry of Multiple Myeloma Adult Patients Treated With Revlimid (Lenalidomide) in China
Brief Title: Observational Registry Study of Chinese Patients Treated With Revlimid (Lenalidomide)
Status: Terminated | Type: Observational
Why Stopped: Business Decision
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: NIPMS-RV-CN-001
Record Dates: First submitted 2013-09-18; First posted 2013-09-20 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Multiple Myeloma
Keywords: Revlimid, lenalidomide, multiple myeloma, PFS, Response Rates
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Multiple Myeloma Patients Treated with Revlimid (lenalidomide): Single Cohort of Multiple Myeloma Patients Treated with Revlimid
  Interventions: Drug: Revlimid (lenalidomide)

INTERVENTIONS:
Drug: Revlimid (lenalidomide) — Revlimid (lenalidomide) as prescribed in usual clinical practice

SUMMARY:
The primary objective of this study is to document efficacy and safety data in a real-world setting of Chinese multiple myeloma patients who have received at least one prior therapy treated with REVLIMID (lenalidomide).

DETAILED DESCRIPTION:
This registry is prospective, multi-center, observational study and will collect efficacy and safety data on multiple myeloma adult patients who have received at least one prior therapy and take REVLIMID as part of standard care associated with patients' treatment in order to characterize the use, efficacy and outcomes of REVLIMID treatment.

The registry will capture data from 600 patients being prescribed REVLIMID in specified hospitals and all patients will be followed in the registry for two years after enrollment of the last patient.

ELIGIBILITY:
Inclusion Criteria:

* Must understand and voluntarily sign written informed consent At least 18 years old at the time of signing informed consent Diagnosed with Multiple Myeloma Must have received at least one prior Multiple Myeloma treatment at the time of signing informed consent

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Chinese Patients with Multiple Myeloma Treated with Revlimid (Lenalidomide) in a Postmarketing setting
Sampling Method: Non-Probability Sample
Enrollment: 176 (Actual)
Dates: Start 2013-11; Primary Completion 2016-07 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | 2 years after enrollment of last patient
  Assessment of PFS using IMWG Uniform Response Criteria
Response Rates | 2 years after enrollment of last patient
  Assessment of Response Rates (CR, VGPR, PR) using IMWG Uniform Response Criteria

SECONDARY OUTCOMES:
Overall Survival (OS) | Two years after last patient enrolled
Time to Response (TTR) and Duration of Response (DOR) | Two years after last patient enrolled
Duration of Treatment with Revlimid | Two years after last patient enrolled.
  Reason for dose interruption/reduction of REVLIMID, if this occurs. Reason for discontinuation of REVLMID
Safety Profile of Revlimid | Two years after last patient enrolled
  All Adverse Events (AEs) and occurrence of second primary malignancies (SPM)

CONTACTS AND LOCATIONS:
Overall Officials: Yu (Flora) Yao, MD, Study Director — Celgene Pharmaceutical (Shanghai) Co. Ltd.
Locations (17):
- China (17):
  - Peking Chao-Yang Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - People's Liberation Army Hospital 307, Beijing
  - Beijing Hospital, Beijing
  - The Fisrt Hospital Of Jilin University, Changchun
  - Xiangya Hospital Central-South University, Changsha
  - Xinqiao Hospital, 3rd Military Medical University, Chongqing
  - NanFang Hospital of China Southern Medical University, Guangzhou
  - The First Affliated Hospital of Anhui Medical University, Hefei
  - Qilu Hospital of Shandong University, Jinan
  - The Affiliated Hospital of Mecical College Qingdao University, Qingdao
  - Shanghai Changzhen Hospital, Shanghai
  - The Second Affiliated Hospital Of China Medical University, Shenyang
  - The First Affiliated Hospital of Suzhou University, Suzhou
  - People's Hospital of Xinjiang Uygur Autonomous Region, Ürümqi
  - Wuhan Union Hospital of Tongji Medical College of Huazhong University of Science & Technology, Wuhan
  - Tongji Medical College Huazhong University of Science & Technology, Wuhan

REFERENCES:
- [Derived] Wang GM, Yang GZ, Huang ZX, Zhong YP, Jin FY, Liao AJ, Wang XM, Fu ZZ, Liu H, Li XL, Zhou JF, Zhang X, Hu Y, Meng FY, Huang XJ, Chen WM, Lu J. [A prospective multi-center trial of non-interventional and observational study of lenalidomide in Chinese patients with multiple myeloma]. Zhonghua Nei Ke Za Zhi. 2017 Jul 1;56(7):500-506. doi: 10.3760/cma.j.issn.0578-1426.2017.07.006. Chinese. PMID 28693058